CLINICAL TRIAL: NCT00369915
Title: The Antidepressant Efficacy of the Anticholinergic Scopolamine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060234; 06-M-0234
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-09

CONDITIONS: Unipolar Depression; Bipolar Depression
Keywords: Cholinergic; Unipolar; Bipolar; Depression; Muscarinic; Scopolamine; Major Depressive Disorder; MDD; Bipolar Disorder; BP
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression; Depressive Disorder, Major | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Plac/Scop (Experimental): Placebo then scopolamine
  Interventions: Drug: Scopolamine
- Scop/Plac (Experimental): Scopolamine then placebo
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Scopolamine
  Arms: Scop/Plac
Drug: Scopolamine
  Arms: Plac/Scop

SUMMARY:
A previous study showed that the intravenous administration of scopolamine produces antidepressant effects. This study is designed to determine if other routes of administration of scopolamine produce antidepressant effects.

DETAILED DESCRIPTION:
Despite the availability of a wide range of antidepressant drugs, clinical trials indicate that 30% to 40% of patients with major depression fail to respond to first-line antidepressant treatment, despite adequate dosage, duration, and compliance. Moreover, in those patients who do experience symptomatic relief following conventional anti-depressant treatment, clinical improvement is not evident for 3-4 weeks. Thus, there is a clear need to develop novel and improved therapeutics for unipolar and bipolar depression.

The cholinergic system is one of the neurotransmitter systems implicated in the pathophysiology of mood disorders. Evidence suggests that during major depressive episodes, the cholinergic system is hypersensitive to acetylcholine. Agents that enhance muscarinic cholinergic receptor function increase depressive symptoms in depressed subjects, and can produce symptoms of depression in healthy individuals. The preclinical literature more specifically implicates the muscarinic receptors and indicates that the use of muscarinic antagonists, in the context of animal models of depression, results in improvement in the behavioral analogs of depression.

Preliminary results obtained under protocol 3-M-0108 provide strong evidence for the potential effectiveness of the anticholinergic scopolamine in rapidly producing clinically significant antidepressant effects. We observed large reductions in Montgomery-Asberg Depression Rating Scale (MADRS) scores that occurred over hours/days following i.v. infusion of scopolamine, which stood in marked contrast to the 3-4 week period generally required for conventional therapies. Moreover, these improvements were observed in subjects who had been nonresponsive or incompletely responsive to conventional antidepressant therapies, highlighting the potential for this treatment to benefit a larger percentage of individuals with depression. The goal of this research project is to perform a clinical trial to evaluate the efficacy of the muscarinic cholinergic receptor antagonist scopolamine administered via transdermal patch on clinical symptoms of depression.

ELIGIBILITY:
* INCLUSION CRITERIA:

Two groups of subjects will be recruited for studies under this protocol: unipolar depressives and bipolar depressives. Subjects with unipolar or bipolar depression appear to exhibit abnormal cholinergic function during the depressed phase, and no differences are hypothesized to exist between MDD and BD depressives herein. However, while BD subjects are more difficult to recruit, the evidence for cholinergic abnormalities has been particularly compelling for BD. Moreover, observations from our pilot study suggest that scopolamine will improve symptoms in both MDD and BD, a particularly persuasive observation given BD notoriously has been difficult to treat. Thus, the magnitude of this serious clinical problem justifies the inclusion of BD subjects. Therefore both groups will be recruited. However, BD Type I subjects will be included only if they are currently stable on lithium or valproate to reduce the risks associated with possible precipitation of mania.

The presence of inclusion and exclusion criteria will be established using both an unstructured clinical interview with a psychiatrist and the Structured Clinical Interview for DSM-IV (SCID). Family history of mental illness will be obtained from the subject using the Family Interview of Genetic Studies. We will recruit 24 subjects per group.

DEPRESSED SAMPLES: Subjects (ages 18-55) currently suffering from a major depressive episode falling into one of the following subgroups:

1. . MAJOR DEPRESSIVE DISORDER (MDD): Subjects will be selected with primary MDD and are currently depressed as defined by DSM-IV criteria for recurrent MDD and current MADRS score in the moderately-to-severely depressed range (greater than or equal to 20). The duration of the index episode is greater than or equal to four weeks.
2. . BIPOLAR DISORDER TYPE II (BD): Subjects will be selected who meet DSM-IV criteria for bipolar disorder Type I or II and are currently depressed, with MADRS score in the moderately-to-severely depressed range (greater than or equal to 20). The duration of the index episode is greater than or equal to four weeks.

EXCLUSION CRITERIA:

Subjects will be recruited who are drug-naive or who have not received psychotropic drugs for at least 3 weeks (8 weeks for fluoxetine) prior to screening. Subjects also will be excluded if they have: a) serious suicidal ideation or behavior, or current delusions or hallucinations, b) inability to provide informed consent, c) serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, endocrinologic, neurologic, immunologic, or hematologic disease, d) a history of drug or alcohol abuse within 6 months or alcohol or drug dependence in the last five years (DSM IV criteria), e) not using a medically accepted means of contraception and are a woman of childbearing potential, f) current pregnancy (documented by pregnancy testing prior to each brain scan to avoid exposing a fetus to radiation or to a research MRI scan that is not medically necessary), g) current breast feeding, h) history of ulcerative colitis or toxic megacolon, i) vision and/or hearing problems severe enough to interfere with testing, j) electrocardiographic evidence of ischemia, arrhythmia, conduction defect, or myocardial infarction, k) current blood pressure of greater than 160 mm Hg or less than 90 mm Hg systolic, or greater than 90 mm Hg diastolic, l) clinically significant cerebrovascular or cardiovascular disease, hypertension, congestive heart disease, angina pectoris, clinic evidence of cerebrovascular disease, gross neurological impairment, hyperthyroidism, known hypersensitivity or idiosyncracy to anticholinergic agents (e.g. skin rashes), glaucoma, renal or hepatic impairment, m) current nicotine use or nicotine dependence within last six months (due to the effects of nicotine on the cholinergic system) n) narrow angle glaucoma (due to the possibility of exacerbation of this condition by scopolamine) o) age greater than 55 years (to reduce the biological heterogeneity encompassed by the MDD and BD criteria, since subjects with a late age-at onset for depression have a far greater likelihood of having MRI correlates of cerebrovascular disease than age-matched, healthy controls or age-matched, early-onset depressives), p) exposure within two weeks to medications likely to affect mood or cognition or likely to interact with scopolamine (e.g. narcotics or anti-cholinergic agents)- as verified by history and urine drug screen, q) HIV positive status, r) history of gastric or intestinal obstructions, s) history of urinary retention or bladder obstruction. During the course of this study, participants will be unable to take some medications, including antidepressant or antianxiety agents, sleep aids, diphenhydramine (e.g. Benedryl) or cough/cold preparations that contain diphenhydramine or antihistamines. A detailed list of allowed and not allowed medications is provided in Appendix B in the protocol.

We are not excluding comorbid anxiety disorders. Exclusion of patients with comorbid anxiety disorders would affect the generalizability of our findings since a substantial percentage of patients with major depression have these comorbid diagnoses. Instead, we will exclude patients with this comorbid diagnosis only if it is believed to be of clinical significance. Allowing participation by patients with histories of comorbid anxiety disorders broadens the inclusion criteria to more closely approximate patients seen in real world settings.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2006-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maura L Furey, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Janowsky DS, el-Yousef MK, Davis JM. Acetylcholine and depression. Psychosom Med. 1974 May-Jun;36(3):248-57. doi: 10.1097/00006842-197405000-00008. No abstract available. PMID 4829619
- [Background] Janowsky DS, el-Yousef MK, Davis JM, Hubbard B, Sekerke HJ. Cholinergic reversal of manic symptoms. Lancet. 1972 Jun 3;1(7762):1236-7. doi: 10.1016/s0140-6736(72)90956-7. No abstract available. PMID 4113219
- [Background] Janowsky EC, Risch C, Janowsky DS. Effects of anesthesia on patients taking psychotropic drugs. J Clin Psychopharmacol. 1981 Jan;1(1):14-20. doi: 10.1097/00004714-198101000-00004. PMID 6117578
- [Derived] Park L, Furey M, Nugent AC, Farmer C, Ellis J, Szczepanik J, Lener MS, Zarate CA Jr. Neurophysiological Changes Associated with Antidepressant Response to Ketamine Not Observed in a Negative Trial of Scopolamine in Major Depressive Disorder. Int J Neuropsychopharmacol. 2019 Jan 1;22(1):10-18. doi: 10.1093/ijnp/pyy051. PMID 30184133
- [Derived] Szczepanik J, Nugent AC, Drevets WC, Khanna A, Zarate CA Jr, Furey ML. Amygdala response to explicit sad face stimuli at baseline predicts antidepressant treatment response to scopolamine in major depressive disorder. Psychiatry Res Neuroimaging. 2016 Aug 30;254:67-73. doi: 10.1016/j.pscychresns.2016.06.005. Epub 2016 Jun 20. PMID 27366831
- [Derived] Drevets WC, Furey ML. Replication of scopolamine's antidepressant efficacy in major depressive disorder: a randomized, placebo-controlled clinical trial. Biol Psychiatry. 2010 Mar 1;67(5):432-8. doi: 10.1016/j.biopsych.2009.11.021. Epub 2010 Jan 15. PMID 20074703

RESULTS

PARTICIPANT FLOW:
Groups:
- Plac/Scop: 6 administrations of placebo patch at 4 to 5 day intervals; followed by 6 administrations of scopolamine patch at 4 to 5 day intervals
- Scop/Plac: 6 administrations of scopolamine patch at 4 to 5 day intervals; followed by 6 administrations of placebo patch at 4 to 5 day intervals
Period: Overall Study
Arm/Group | Plac/Scop | Scop/Plac
Started | 10 | 7
Completed | 4 | 4
Not Completed | 6 | 3
Not completed — expected side effects | 2 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — W/drawl by investigators | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plac/Scop | Scop/Plac | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6.6) | 33 (10.4) | 31.9 (8.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Severity
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) has a range of scores from 0 to 60 where the highest values indicate the most depression.
Time Frame: Outcome measures obtained at each of 12 sessions
Population: Only participants who completed the trial were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plac/Scop | Scop/Plac
Number analyzed (Participants) | 4 | 4
units on a scale
  Block 1 - Session 1 | 29.5 (2.5) | 30.5 (4.2)
  Block 1 - Session 2 | 26.5 (8.2) | 29.8 (1.5)
  Block 1 - Session 3 | 24.5 (3.7) | 31.0 (2.9)
  Block 1 - Session 4 | 19.5 (6.6) | 27.0 (5.5)
  Block 1 - Session 5 | 19.3 (7.4) | 27.8 (5.6)
  Block 1 - Session 6 | 20.8 (4.5) | 28.5 (6.2)
  Block 2 - Session 1 | 23.3 (3.7) | 27.5 (7.9)
  Block 2 - Session 2 | 18.0 (3.8) | 23.8 (6.7)
  Block 2 - Session 3 | 19.8 (8.3) | 20.0 (6.5)
  Block 2 - Session 4 | 18 (9.1) | 17.3 (9.1)
  Block 2 - Session 5 | 16.3 (7.9) | 16.8 (9.7)
  Block 2 - Session 6 | 15.5 (8.8) | 20.3 (9.3)

2. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale (HARS) has a range of scores from 0 to 56 where the highest values indicate the most anxiety.
Time Frame: Each of 12 sessions.
Population: Only study completers were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plac/Scop | Scop/Plac
Number analyzed (Participants) | 4 | 4
units on a scale
  Block 1 - Session 1 | 17.0 (6.2) | 20.3 (9.0)
  Block 1 - Session 2 | 16.8 (6.2) | 14.5 (2.7)
  Block 1 - Session 3 | 14.5 (8.4) | 14.3 (4.7)
  Block 1 - Session 4 | 14.3 (6.5) | 13.0 (2.8)
  Block 1 - Session 5 | 12.8 (5.0) | 12.0 (4.7)
  Block 1 - Session 6 | 17.8 (7.1) | 11.5 (5.3)
  Block 2 - Session 1 | 14.8 (2.2) | 13.5 (7.9)
  Block 2 - Session 2 | 13.3 (3.8) | 12.0 (7.6)
  Block 2 - Session 3 | 14.3 (4.0) | 13.3 (5.6)
  Block 2 - Session 4 | 10.5 (2.7) | 14.3 (9.0)
  Block 2 - Session 5 | 9.8 (2.1) | 10.3 (6.0)
  Block 2 - Session 6 | 11.8 (3.2) | 11.8 (6.9)

ADVERSE EVENTS:
Arm/Group | Plac/Scop | Scop/Plac
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 2/10 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plac/Scop (N=10) | Scop/Plac (N=7)
mild confusion (Psychiatric disorders) | 1 (1) | 1 (1)
dry mouth (Psychiatric disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes